CLINICAL TRIAL: NCT06357624
Title: Effectiveness of Mulligan Mobilization Technique in Individuals With Non-spesific Neck Pain
Brief Title: Effectiveness of Mulligan Mobilization Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Tarik Ozmen, Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physiotherapy
Record Dates: First submitted 2024-03-10; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Neck Pain; Disability Physical; Kinesiophobia
MeSH Terms: conditions — Neck Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan mobilization technique (Experimental): The participants received MMT from the physiotherapist.
  Interventions: Other: Mulligan mobilization; Other: Self-Mobilization
- Self-mobilization techniques (Other): The second group was trained only self-mobilization technique.
  Interventions: Other: Self-Mobilization

INTERVENTIONS:
Other: Mulligan mobilization — The SNAGS technique was applied to 3 sets of 10 repetitions with 15-30 seconds rest between sets while the participants were in a sitting position. A physiotherapist applied passive motion to facet joints at each spinal level. The participant was questioned in which direction he/she felt pain during cervical ROM and the application was carried out in the painful/limited directions.
  Arms: Mulligan mobilization technique
Other: Self-Mobilization — For the self-mobilization technique, each participant was asked to extend a pain-free while pushing upwards from the transverse processes of the treated vertebra with the thumbs of both hands. In addition, the middle or index finger of the right hand was asked to pull the treated vertebra to the right side, while at the same time, left rotation was asked at the pain limit. Self-mobilization was applied every day, twice a day, five times.

SUMMARY:
The aim of this study was to investigate the effects of the Mulligan mobilization technique (MMT) on pain intensity, joint position sense (JPS), kinesiophobia, and disability level in individuals with nonspecific neck pain. A total of 34 female individuals with nonspecific neck pain were included in the study. Pain intensity, JPS, kinesiophobia, and disability levels of all participants were evaluated before and after the 3-week intervention. Participants were randomly divided into two groups. In the first group, the participants received MMT by the physiotherapist twice a week for 3 weeks, and self-mobilization techniques as a home exercise program. The second group was trained only self-mobilization techniques.

DETAILED DESCRIPTION:
A total of 34 female individuals with nonspecific neck pain that persisted for at least 3 months were included in the study. Individuals who had a surgical indication for the cervical region and/or had undergone surgery, who had received physiotherapy or other treatment in the last year due to neck pain, who had a history of trauma to the cervical and thoracic region, and who additionally had a musculoskeletal system disease were excluded. All participants were evaluated for pain intensity, JPS, kinesiophobia, and disability levels before and after the 3-week intervention. Participants were randomly divided into two groups using the coin toss method. In the first group, the participants received MMT by the physiotherapist twice a week for 3 weeks, and self-mobilization techniques as a home exercise program. The second group was trained only self-mobilization technique.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific neck pain

Exclusion Criteria:

* History of trauma to the cervical and thoracic region

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Disability | Three weeks
  The Neck Disability Index (NDI) was used to determine the severity of disability.It consists of 10 items related to subjective symptoms and activities of daily living. Each item is scored from 0 to 5 points. The total score of the NDI ranges from 0 to 50 points. A higher total score indicates a higher level of disability.
Neck Pain Severity | Three weeks
  Neck Pain intensity was evaluated with Visual Analogue Scale.Pain intensity was evaluated with Visual Analogue Scale (VAS). Participants were asked to mark the intensity of pain they felt on a 100 mm long horizontal line marked "0" at one end and "10" at the other. "0" indicates no pain, and "10" indicates very severe pain.
Joint Position Sense | Three weeks
  Cervical JPS was measured by using CROM

CONTACTS AND LOCATIONS:
Locations (1):
- Tarik Ozmen, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alansari SM, Youssef EF, Shanb AA. Efficacy of manual therapy on psychological status and pain in patients with neck pain. A randomized clinical trial. Saudi Med J. 2021 Jan;42(1):82-90. doi: 10.15537/smj.2021.1.25589. PMID 33399175
- [Background] Buyukturan O, Buyukturan B, Sas S, Kararti C, Ceylan I. The Effect of Mulligan Mobilization Technique in Older Adults with Neck Pain: A Randomized Controlled, Double-Blind Study. Pain Res Manag. 2018 May 15;2018:2856375. doi: 10.1155/2018/2856375. eCollection 2018. PMID 29861800
- [Background] Ganesh GS, Mohanty P, Pattnaik M, Mishra C. Effectiveness of mobilization therapy and exercises in mechanical neck pain. Physiother Theory Pract. 2015 Feb;31(2):99-106. doi: 10.3109/09593985.2014.963904. Epub 2014 Sep 29. PMID 25264016